CLINICAL TRIAL: NCT03876587
Title: A Multicenter, Phase II Open Label Study of Pyrotinib Maleate Combined With Docetaxel in the First-line Treatment of HER2-positive Metastatic Breast Cancer
Brief Title: Pyrotinib Combined With Docetaxel in the First-line Treatment of HER2-positive MBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaojia Wang(xj wang), Director, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-001
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Pyrotinib Maleate; HER2 Targeted Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Pyrotinib Maleate combine with Docetaxel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Maleate combine with Docetaxel (Experimental): Pyrotinib Maleate combine with Docetaxel should be administrate to all subjects.
  Initial dose: Pyrotinib Maleate 400mg oral administration everyday plus Docetaxel 75mg per square of BSA every three weeks intravenous injection.
  Interventions: Drug: Pyrotinib Maleate combine with Docetaxel

INTERVENTIONS:
Drug: Pyrotinib Maleate combine with Docetaxel — Pyrotinib Maleate combine with Docetaxel as the first-line treatment to HER2-positive Metastatic Breast Cancer

SUMMARY:
To explore the efficacy and safety of pyrotinib combined with docetaxel regimen in the first-line treatment of HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
A multi-center, one-arm, open label design study,which is planned to enroll 79 patients with HER2-positive metastatic breast cancer receiving first-line treatment with pyrotinib and docetaxel. The main purpose of this study was to observe the efficacy and safety of first-line treatment with pyrrolidine and docetaxel for HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Local recurrent or metastatic breast cancer suitable for chemotherapy, confirmed histologically.
* HER2-positive breast cancer(according to 2018 ASCO/CAP HER2 test guideline).
* do not chemotherapy for recurrent and metastatic lesions, but local treatment for local symptoms, such as radiotherapy for relieving bone pain, is allowed.
* if the patient is bilateral breast cancer, metastasis lesions must be HER2-positive.
* 18-70 years old.
* ECOG PS 0～1.
* life expectancy is not less than 12 weeks.
* at least one measurable lesion according to RECIST 1.1.
* Endocrine therapy is allowed to relapse/metastasis disease; patients with previous adjuvant/neoadjuvant use of Taxus and trastuzumab, disease-free interval from the end of last adjuvant/neoadjuvant Taxus therapy to the progression of tumors (≥12 months), and disease-free interval from the end of last adjuvant/neoadjuvant trastuzumab to the progression of tumors (≥ 6 months).
* ANC ≥ 1.5×109/L,PLT ≥ 75×109/L,Hb ≥ 100 g/L;TBIL≤1.0ULN；ALT and AST≤3×ULN（ALT and AST≤5×ULN if liver metastasis）;BUN and Cr≤1.5×ULN and CCr≥50 mL/min.
* LVEF ≥ 50% and QTc≤480 ms.
* known hormone receptor status.
* Signed informed

Exclusion Criteria:

* Central nervous system metastasis.
* Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption.
* patient who received radiotherapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks before admission; those who received anti-tumor endocrine therapy after screening period
* Participated in other drug clinical trials within 4 weeks before admission
* Tyrosine kinase inhibitors targeting HER2 (Neratinib, Lapatinib, pyrotinib, etc.) have been used or are being used in the past.
* Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.
* Receive other antitumour treatment at the same time
* A history of immunodeficiency, including HIV positive, HCV, active hepatitis B, or other acquired, congenital immunodeficiency disorders, or organ transplantation, is known.
* Has suffered from any heart disease
* Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial
* According to the judgement of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of research (including, but not limited to, severe hypertension, severe diabetes, active infections, etc.).
* The patient did not recover from the toxicity of previous treatment to grade 0-1 (except hair loss).
* History of neurological or psychiatric disorders
* Along with CYP3A4 inhibitors or inducers or drugs that are using to prolong the QT interval
* Researchers believe that patients are not suitable for any other situation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | from enrollment to progression or death (for any reason), assessed up to 100 months
  Ratio of CR and PR in all subjects

SECONDARY OUTCOMES:
PFS | from enrollment to progression or death (for any reason),assessed up to 100 months
  Progression-Free Survival
DoR | The first evaluation of CR or PR to progression or death (for any reason),assessed up to 100 months
  Duration of Response
Clinical Benefit Rate | from enrollment to progression or death (for any reason),assessed up to 100 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects
OS | from enrollment to death (for any reason).assessed up to 100 months
  Overall Survival

OTHER OUTCOMES:
adverse event | from enrollment to 30 days after the last dose administrate
  Adverse events are described in terms of CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, chief doctor, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
the data will be shared from the trial begin and for 10 years.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: from the trial begin and for 10 years.
Access Criteria: every one

REFERENCES:
- [Derived] Dai L, Gao T, Guo R, Chen Y, Wang J, Zhou S, Tang Y, Chen D, Huang S. Efficacy and safety of pyrotinib-based regimens in HER2 positive metastatic breast cancer: A retrospective real-world data study. Neoplasia. 2024 Oct;56:101029. doi: 10.1016/j.neo.2024.101029. Epub 2024 Jul 17. PMID 39024777
- [Derived] Zheng Y, Cao WM, Shao X, Shi Y, Cai L, Chen W, Liu J, Shen P, Chen Y, Wang X, Li H, Li M, Chen Z, Wang X. Pyrotinib plus docetaxel as first-line treatment for HER2-positive metastatic breast cancer: the PANDORA phase II trial. Nat Commun. 2023 Dec 14;14(1):8314. doi: 10.1038/s41467-023-44140-y. PMID 38097605